CLINICAL TRIAL: NCT05129384
Title: Colonization of the Infant Gut With B. Infantis EVC001 to Reduce Symptoms of Colic
Brief Title: The COLIC Study: Colonization of the Infant Gut With B. Infantis EVC001 to Reduce Symptoms of Colic
Acronym: COLIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company pursuing other research paths
Sponsor: Evolve BioSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EV-9101
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-06

CONDITIONS: Infantile Colic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Intervention Model Description: Infants will be randomized 1:1 to one of two study arms (treatment or placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind, randomized, placebo-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): B. infantis EVC001 infant probiotic
  Interventions: Dietary Supplement: B. infantis EVC001 or Lactose Placebo
- Placebo (Placebo Comparator): Lactose
  Interventions: Dietary Supplement: B. infantis EVC001 or Lactose Placebo

INTERVENTIONS:
Dietary Supplement: B. infantis EVC001 or Lactose Placebo — Infant probiotic
  Other Names: Lactose Placebo

SUMMARY:
To investigate whether B. infantis EVC001 colonization in the infant gut can reduce symptoms of colic

DETAILED DESCRIPTION:
There is evidence to support that B. infantis EVC001 supplementation may ameliorate symptoms associated with colic by establishing and maintaining the necessary gut microbial composition to promote proper barrier and immune function in infants. The primary objective of this study is to assess the effect of the probiotic, B. infantis EVC001, on reducing the duration of crying/fussing symptoms of breastfed infants diagnosed with infantile colic from Baseline to Day 14.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a diagnosis of infantile colic per Rome IV criteria and reported to cry/fuss for ≥ 3 hours/day, within a 24-hour period as determined by the 24-hour cry/fuss eDiary AND 24 hours of LENA vocalizations
* Infants with a gestational period of ≥ 37 to 42 weeks
* Infants between 14 and ≤ 42 days of life at the completion of screening/baseline tasks
* Infants exclusively breastfed for at least 7 days immediately prior to enrollment and with mother's intent to continue feeding breast milk exclusively for the duration of the study
* Mothers willing to use their own electronic device(s) to download and utilize all required study software (decentralized trial platform on a mobile device and the LENA device software on a Windows 10 or higher laptop or desktop that has at least 10 GB of free space and fast, reliable internet)
* Mother is fluent in English

Exclusion Criteria:

* Infants born in multiple birth (i.e., twins, triplets, etc.)
* Infants born with medical complications (i.e., neurological, cerebral palsy, confirmed food allergies)
* Infants with current evidence of failure to thrive, fever, or illness
* Infants with any GI tract abnormalities
* Antibiotic, infant formula, solid food or iron supplement intake within 7 days prior to enrollment or mother's intent to feed non-study probiotics, prebiotics, infant formula, solid food or iron supplements to their infant at any time during the study
* Infants who have consumed any probiotics since birth
* Unwillingness to discontinue/avoid products used to treat IC (i.e., Simethicone, gripe water, colic drops, etc.) during the study. Note: consumption of IC products prior to the baseline period is NOT exclusionary
* Maternal use of probiotics containing B. infantis during pregnancy, after the baby's birth and/or intent to use probiotics containing B. infantis at any time throughout the study
* Maternal smoking or smoking within the home by any household member currently or during pregnancy
* Mother following exclusionary diet due to her infant's colic (i.e., dairy elimination diet)
* Any infant the Investigator deems to be ineligible for participation

Ages: 14 Days to 42 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in crying/fussing duration | Baseline to Day 14
  Assess the effect of the probiotic, B. infantis EVC001, on duration of crying/fussing symptoms of breastfed infants diagnosed with infantile colic

CONTACTS AND LOCATIONS:
Overall Officials: Robin Flannery, Study Director — Evolve BioSystems; Parth Shah, Principal Investigator — Obvio Health
Locations (1):
- Obvio Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Our intent is to share group/averaged data for the cohorts to decrease risks associated with patient anonymity